CLINICAL TRIAL: NCT02500901
Title: Combined Targeting of the Androgen Receptor in Metastatic Castrate-Resistant Prostate Cancer With Enzalutamide and the Poly (ADP- Ribose) Polymerase (PARP) Inhibitor Niraparib: Hoosier Cancer Research Network GU14-202
Brief Title: Enzalutamide and Niraparib in the Treatment of Metastatic Castrate-Resistant Prostate Cancer (CRPC)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Suspended by funder
Sponsor: Paul Mathew, MD (Other)
Collaborators: Hoosier Cancer Research Network (Other); Tesaro, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Paul Mathew, MD, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCRN GU14-202
Record Dates: First submitted 2015-07-02; First posted 2015-07-17 (Estimated); Results first posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Metastatic Prostate Cancer
Keywords: Enzalutamide; Niraparib; PARP-1 inhibitor; PARP-2 inhibitor; Castrate-Resistant Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental Treatment (Experimental): Subjects will receive enzalutamide 160 mg/day PO in a 28-day lead-in cycle to assess tolerability. If well-tolerated, cycle 1 of combined enzalutamide and niraparib will commence. Enzalutamide will continue at 160 mg PO daily. Niraparib will be administered in three dose-escalation cohorts of 100mg PO, 200mg PO or 300 mg PO daily. Six subjects will be enrolled at each dose level. Each cycle will be 28 days. Combination treatment will continue until documented progression, unmanageable toxicity, or subject or treating investigator decision to discontinue for any reason.
  Interventions: Drug: Enzalutamide; Drug: Niraparib

INTERVENTIONS:
Drug: Enzalutamide — Following completion of 28-day lead-in cycle, enzalutamide 160 mg PO daily will continue to be administered in 28-day cycles until documented progression, unmanageable toxicity, or decision to discontinue for any reason.
  Other Names: Xtandi
Drug: Niraparib — Niraparib will be administered daily in three dose-escalation cohorts of 6 subjects per dose levels of 100mg PO, 200mg PO or 300mg PO in 28-day cycles until documented progression, unmanageable toxicity, or decision to discontinue for any reason.

SUMMARY:
This is a phase I study to determine the safety and feasibility of the combination of enzalutamide and niraparib in subjects with metastatic castration-resistant prostate cancer (CRPC).

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center trial.

INVESTIGATIONAL TREATMENT:

Each eligible subject will begin treatment with a 28-day enzalutamide 160 mg/day lead-in cycle. If a subject is able to tolerate the lead-in enzalutamide cycle without Grade 2 or Grade 2-4 drug-related toxicity, dose reduction, or missed doses due to toxicity, cycle 1 of combined enzalutamide and niraparib will commence. Enzalutamide will continue at 160 mg daily.

Niraparib will be dosed daily starting at 100mg (dose level 1). Six subjects will be enrolled per dose level. If less than 33% of the subjects experience a dose-limiting toxicity (DLT) at the beginning of cycle 2, then the daily dose of niraparib will escalate to 200mg (dose level 2). If dose level 2 is similarly tolerated, then the daily dose of niraparib escalate to 300mg (dose level 3).

The following required laboratory values must be obtained within 14 days prior to registration for protocol therapy:

Hematopoietic:

* White blood cell count (WBC) ≥ 1500/mm3
* Hemoglobin (Hgb) ≥ 9 g/dL
* Platelets ≥ 150,000/µL
* Absolute neutrophil count (ANC) ≥ 1500/mm3

Renal:

* Calculated creatinine clearance of ≥ 40 cc/min using the Cockcroft-Gault formula

Hepatic:

* Bilirubin ≤ 1.5 × upper limit of normal (ULN)
* Aspartate aminotransferase (AST, SGOT) ≤ 2.5 × ULN

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Age ≥ 18 years at the time of consent.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1 within 14 days prior to registration.
* Men who are not surgically sterile (vasectomy) must agree to use an acceptable method of contraception. Male subjects with female sexual partners who are pregnant, possibly pregnant, or who could become pregnant during the study must agree to use condoms from the first dose of study drug through at least 120 days after the last dose of study drug. Total abstinence for the same study period is an acceptable alternative.
* Documented histologically or cytologically confirmed adenocarcinoma of the prostate.
* Ongoing androgen deprivation therapy with a Gonadotropin Releasing Hormone (GnRH) analogue or bilateral orchiectomy. Subjects who have not undergone orchiectomy must plan to continue GnRH analogue therapy for the duration of the trial.
* All subjects on oral anti-androgen therapy must have been off therapy for at least 4 weeks prior to registration (6 weeks for bicalutamide) to exclude an anti-androgen withdrawal response. Patients who received secondary anti-androgen therapy and did not exhibit a >50% PSA decline, or subjects with any rise in PSA, objective or symptomatic progression following anti-androgen withdrawal will not be required to meet this withdrawal requirement.
* Documented metastatic disease with prostate-specific antigen (PSA) progression, radiographic progression, or both, despite receiving luteinizing hormone releasing hormone (LHRH) analogue therapy or orchiectomy with a serum testosterone level of 50 ng/dL or less.

  * PSA progression is defined as three successive rising PSA values with an interval of at least one week between determinations.
  * Radiographic progression is defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria or at least two new lesions on bone scan.
* At screening the serum testosterone must be 50 ng/dL or less and the PSA must be greater or equal to 2 ng/mL.
* Estimated life expectancy > 6 months
* Prior treatment of CRPC, including docetaxel, cabazitaxel, sipuleucel-T, or Radium-223 is allowed.
* Prior therapy with abiraterone allowed for a maximum of 9 subjects.
* Prior chemotherapy must be completed at least 28 days prior to registration and the participant subject must have recovered from the acute toxic effects.

Exclusion Criteria:

* Prior enzalutamide or other next-generation androgen receptor- (AR) targeting therapy.
* Prior PARP-inhibitor therapy.
* History of or active central nervous system (CNS) metastases. Subjects with neurological symptoms must undergo a head computed tomography (CT) scan or brain magnetic resonance imaging (MRI) to exclude brain metastasis.
* Radioisotope or external beam radiation exposure in the last 4 weeks. Exposure to strontium, regardless of when exposure occurred.
* Prior radiation to 25% or more of the bone marrow.
* Treatment with any investigational agent within 28 days prior to registration.
* Known significant immunodeficiency as determined by the site investigator.
* Prior malignancy except for adequately treated basal cell or squamous cell skin cancer, or other cancer for which the subject has been disease-free or stable for at least one year.
* Prolonged QTc over 470 ms.
* History of seizure.
* Clinically significant active infections on systemic therapy as judged by the site investigator.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-03; Primary Completion 2016-05-10 (Actual); Study Completion 2016-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Mathew, M.D., Study Chair — Hoosier Cancer Research Network
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Hoosier Cancer Research Network Website — http://www.hoosieroncologygroup.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Treatment: enzalutamide 160 mg/day PO in a 28-day lead-in cycle to assess tolerability. If well-tolerated, cycle 1 of combined enzalutamide and niraparib will commence. Enzalutamide will continue at 160 mg PO daily. Niraparib will be administered in three dose-escalation cohorts of 100mg PO, 200mg PO or 300 mg PO daily. Six subjects will be enrolled at each dose level. Each cycle will be 28 days. Combination treatment will continue until documented progression, unmanageable toxicity, or subject or treating investigator decision to discontinue for any reason.
  Enzalutamide: Following completion of 28-day lead-in cycle, enzalutamide 160 mg PO daily will continue to be administered in 28-day cycles until documented progression, unmanageable toxicity, or decision to discontinue for any reason.
  Niraparib: Niraparib will be administered daily in three dose-escalation cohorts of 6 subjects per dose levels of 100mg PO, 200mg PO or 300mg PO in 28-day cycles until documented
Period: Overall Study
Arm/Group | Experimental Treatment
Started | 2
Completed | 0
Not Completed | 2
Not completed — Disease ProgressionDD | 2

BASELINE CHARACTERISTICS:
Arm/Group | Experimental Treatment
Number analyzed (Participants) | 2
Age, Continuous [Mean (Full Range); unit: years] | 77 [75 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2
Eastern Cooperative Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) from 0-5 that describes a patient's level of functioning where 0=Fully active, able to carry on all pre-disease performance without restriction and 5=Dead:
  Participants
    ECOG 0 | 1
    ECOG 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) for Subjects Receiving Enzalutamide With Niraparib Without Experiencing Dose-limiting Toxicity(s) (DLT)
Description: MTD of niraparib in combination with enzalutamide and MTD for phase II testing.
Time Frame: From the start of combination treatment D29 until 30 days after last dose of study treatment per CTCAE v4, assessed up to 52 weeks
Population: Sufficient data was not collected to determine the maximum tolerated dose (MTD) before study termination.
Arm/Group | Experimental Treatment
Number analyzed (Participants) | 0

2. Secondary Outcome: Progression-free Survival (PFS) With Enzalutamide and Niraparib Combination Therapy.
Description: PFS per RECIST v1.1 for subjects on this combination therapy.
Time Frame: From the date of enrollment until the criteria for disease progression is met as defined by RECIST 1.1 or death from any cause, whichever occurs first, assessed up to 52 weeks
Population: Sufficient data was not collected or analyzed for this secondary objective before study termination.
Arm/Group | Experimental Treatment
Number analyzed (Participants) | 0

3. Secondary Outcome: Objective Response (OR) Rates for All Subjects With Confirmed Partial Response (PR) or Complete Response (CR) Outcomes, Per RECIST v1.1
Description: OR outcomes for subjects on this combination therapy, per RECIST v1.1
Time Frame: From the date of enrollment until the date of documented disease progression or the date of death from any cause, whichever occurs first, assessed up to 52 weeks
Population: Sufficient data was not collected or analyzed for this secondary objective before study termination.
Arm/Group | Experimental Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Duration of participation in study, or until disease progression, up to 24 months.
Arm/Group | Experimental Treatment
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Treatment (N=2)
FALL (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Treatment (N=2)
ANEMIA (Blood and lymphatic system disorders) | 1 (5)
BUTTOCK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 2 (2)
CREATININE INCREASED (Investigations) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 2 (4)
DIZZINESS (Nervous system disorders) | 1 (2)
DRY MOUTH (Gastrointestinal disorders) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 1 (3)
EDEMA LIMBS (General disorders) | 2 (3)
FATIGUE (General disorders) | 2 (3)
HEADACHE (Nervous system disorders) | 1 (2)
HYPERTENSION (Vascular disorders) | 1 (1)
HYPERURICEMIA (Metabolism and nutrition disorders) | 1 (1)
MEMORY IMPAIRMENT (Nervous system disorders) | 1 (1)
NAIL DISCOLORATION (Skin and subcutaneous tissue disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1 (1)
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 (1)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 (1)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (Skin and subcutaneous tissue disorders) | 1 (1)
THROMBOEMBOLIC EVENT (Vascular disorders) | 1 (1)
URINARY INCONTINENCE (Renal and urinary disorders) | 1 (1)
WEIGHT LOSS (Investigations) | 1 (1)
WHITE BLOOD CELL DECREASED (Investigations) | 1 (2)

LIMITATIONS AND CAVEATS:
Study was terminated early by the funder.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No